CLINICAL TRIAL: NCT00712634
Title: A Phase I Dose Escalation Study of Lipopeptide Vaccines With Activity Against Human Cytomegalovirus
Brief Title: Cytomegalovirus Vaccine in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Don Diamond, City of Hope Comprehensive Cancer Center
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000599675; P01CA030206 (NIH); CHNMC-97092
Record Dates: First submitted 2008-07-09; First posted 2008-07-10 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-12

CONDITIONS: Precancerous/Nonmalignant Condition
Keywords: cytomegalovirus infection
MeSH Terms: conditions — Precancerous Conditions; Cytomegalovirus Infections

ARMS (2):
- CMV-seropositive participants (Experimental): Participants are randomized to receive 1 of 4 escalating doses of CMVpp65-A*0201 peptide vaccine containing either helper T-lymphocyte (HTL) PADRE peptide or HTL tetanus toxoid peptide. Within each vaccine dose group, two participants are randomized to receive a placebo. Participants receive the vaccine or a placebo subcutaneously (SC) on days 0 and 28 in the absence of unacceptable toxicity.
  Interventions: Biological: CMVpp65-A*0201 peptide vaccine
- CMV-seronegative participants (Experimental): Participants are randomized to receive 1 of 4 established doses (established in CMV-seropositive participants) of CMVpp65-A*0201 peptide vaccine containing either HTL PADRE peptide or HTL tetanus toxoid peptide. Participants receive the vaccine on days 0, 28, and 56 in the absence of unacceptable toxicity. Participants with a partial or low-level immune response receive one additional booster vaccine on day 90.
  Interventions: Biological: CMVpp65-A*0201 peptide vaccine

INTERVENTIONS:
Biological: CMVpp65-A*0201 peptide vaccine — Vaccine received on either days 0 and 28 or on days 0, 28, and 56 and perhaps day 90

SUMMARY:
RATIONALE: Vaccines may help the body build an effective immune response against cytomegalovirus.

PURPOSE: This randomized phase I trial is studying the side effects and best dose of cytomegalovirus vaccine in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* To establish whether 4 dose levels of the CMVpp65-A*0201 peptide vaccine are safe and well tolerated in cytomegalovirus (CMV)-seropositive participants.
* To determine whether the CMVpp65-A*0201 peptide vaccine, when given as a single injection followed by one booster injection at a safe and well-tolerated dose, is capable of stimulating a memory response in CMV-seropositive participants.
* To evaluate whether CMV-seronegative participants generate a de novo immune response against CMV after immunization with CMVpp65-A*0201 peptide vaccine given as a single injection followed by three booster injections.
* To determine the duration of immune enhancement of CMV-specific cytotoxic T-lymphocyte function as assessed for up to 12 months after primary or secondary immunization with the CMVpp65-A*0201 peptide vaccine.

OUTLINE: This is a dose-escalation study of CMVpp65-A*0201 peptide vaccine in cytomegalovirus (CMV)-seropositive participants. Once a safe dose is established, CMV-seronegative participants are accrued and immunized at that dose. Participants are stratified according to gender.

* CMV-seropositive participants: Participants are randomized to receive 1 of 4 escalating doses of CMVpp65-A*0201 peptide vaccine containing either helper T-lymphocyte (HTL) PADRE peptide or HTL tetanus toxoid peptide. Within each vaccine dose group, two participants are randomized to receive a placebo. Participants receive the vaccine or a placebo subcutaneously (SC) on days 0 and 28 in the absence of unacceptable toxicity.
* CMV-seronegative participants: Participants are randomized to receive 1 of 4 established doses (established in CMV-seropositive participants) of CMVpp65-A*0201 peptide vaccine containing either HTL PADRE peptide or HTL tetanus toxoid peptide. Participants receive the vaccine on days 0, 28, and 56 in the absence of unacceptable toxicity. Participants with a partial or low-level immune response receive one additional booster vaccine on day 90.

Participants undergo blood sample collection at baseline and periodically during study for immunologic laboratory studies. Participants also undergo skin biopsy at baseline. Laboratory studies include assessment of human cytotoxic T-lymphocyte activity and response by ^51chromium-release assay, limiting-dilution analysis, and T-cell proliferation assay; and CD4/CD8 phenotyping by FACScan® flow cytometry.

After completion of study therapy, participants are followed for 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participant
* Cytomegalovirus seropositive or seronegative
* HLA-A*0201-positive

PATIENT CHARACTERISTICS:

* CBC within 1.5 times normal
* SMA-18 within 1.5 times normal
* Hepatitis B virus antigen seronegative
* Hepatitis C virus seronegative
* No diagnosis that is associated with immunodeficiency, including HIV infection
* No serious abnormalities by EKG (in participants ≥ 50 years of age)
* Not pregnant

PRIOR CONCURRENT THERAPY:

* More than 6 months since prior surgery
* No concurrent daily medications for chronic or current illness, except for the following:

  * Thyroid replacement therapy
  * Estrogen replacement therapy
  * Dietary vitamins and protein supplements
  * Antihistamine medication
  * Anticholesterol medication
  * Cardiac and antihypertensive medication
  * Any medication, as determined by the principal investigator, that is not known or likely to be immunosuppressive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 1997-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity
Immunologic response
Duration of immunologic response

CONTACTS AND LOCATIONS:
Overall Officials: Don Diamond, PhD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States